CLINICAL TRIAL: NCT02504944
Title: Safety and Efficacy of Propranolol 0.2% Eye Drops in Treating Newborn With Retinopathy of Premature: A Pilot Study (DROP-ROP-0.2%)
Brief Title: Safety and Efficacy of Propranolol 0.2% Eye Drops in Treating Retinopathy of Premature: A Pilot Study (DROP-ROP-0.2%)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Luca Filippi, MD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DROP-ROP-0.2%
Record Dates: First submitted 2015-07-19; First posted 2015-07-22 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of prematurity; Propranolol; Newborn; Eye Drops; Retinal angiogenesis; Retinal neovascularization
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Neovascularization | interventions — Propranolol; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propranolol 0.2% eye drops (Experimental): Enrolled preterm newborns will receive propranolol as ophthalmic solution (0.2%). The treatment will be started as soon as the diagnosis of stage 1 ROP is made and will be continue until the development of retinal vascularization is completed, but no more than 90 days. Cardiovascular and respiratory parameters will be continuously monitored. Blood samplings checking metabolic, renal and liver functions will be performed periodically, as well as cardiac function, in order to verify the treatment safety. Propranolol concentrations will be measured on dried blood spots at the steady state (10th day). Serial ophthalmological evaluations will be planned to monitor the efficacy of the treatment, the ROP progression and the possible complications.
  Interventions: Drug: Propranolol 0.2% eye drops

INTERVENTIONS:
Drug: Propranolol 0.2% eye drops — Enrolled preterm newborns will receive propranolol as ophthalmic solution (0.2%): 3 microdrops of 6 microliters (μL) propranolol solution (= 6 μg propranolol/microdrop) will be topically applied with a calibrated pipette, in each eye, four times daily (every 6 hours). Propranolol treatment will be always associated to the conventional approach adopted by the Early Treatment for Retinopathy of Prematurity Study (ETROP) Cooperative Group.

SUMMARY:
The aim of the present study is to evaluate the safety and efficacy of propranolol 0.2% eye drops in treating preterm newborns with a precocious stage of retinopathy of prematurity (ROP). Preterm newborns (gestational age 23-32 weeks) with a stage 1 ROP will receive propranolol 0.2% eye drops treatment until retinal vascularization will be completed, but no more than 90 days.

Propranolol concentrations will be measured on dried blood spots at the steady state (10th day). Cardiovascular and respiratory parameters will be continuously monitored. Blood samplings checking metabolic, renal and liver functions will be performed periodically, as well as cardiac function, in order to verify the treatment safety. Serial ophthalmological evaluations will be planned to monitor the efficacy of the treatment, the ROP progression and the possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (gestational age 23-32 weeks) with stage 1 ROP
* A signed parental informed consent

Exclusion Criteria:

* Newborns with heart failure
* Newborns with recurrent bradycardia (heart rate < 90 beat per minute)
* Newborns with second or third degree atrioventricular block
* Newborns with congenital cardiovascular anomalies, except for persistent ductus arteriosus, patent foramen ovale and small ventricular septal defects
* Newborns with hypotension
* Newborns with renal failure
* Newborns with actual cerebral haemorrhage
* Newborns with other diseases which contraindicate the use of beta-adrenoreceptor blockers.
* Newborns with a more severe stage of ROP than stage 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Incidence rate of progression from stage 1 ROP to zone II stage 2 ROP with plus | participants will be followed for the duration of hospital stay, an expected average of 2 months
Incidence rate of progression from stage 1 ROP to zone II stage 3 ROP with plus | participants will be followed for the duration of hospital stay, an expected average of 2 months
Plasma concentrations of propranolol at the steady state measured by dried blood spots | 10th day of treatment

SECONDARY OUTCOMES:
Number of newborns who progress to Stage 2 without plus ROP | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who progress to Stage 3 without plus ROP | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who progress to Stage 4 with total or partial retinal detachment | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who progress to Stage 5 ROP with total or partial retinal detachment | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who need vitrectomy | participants will be followed for the duration of hospital stay, an expected average of 2 months
Collection of adverse events due to eye drop propranolol treatment | participants will be followed for the duration of hospital stay, an expected average of 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Luca Filippi, MD, Principal Investigator — A. Meyer University Childrens' Hospital
Locations (7):
- Italy (7):
  - Neonatal Intensive Care Unit, Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Neonatal Intensive Care Unit, A. Meyer University Childrens' Hospital, Florence
  - Institute of Pediatrics and Neonatology, Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, University of Milan, Milan
  - Neonatal Intensive Care Unit, Azienda Ospedaliera San Gerardo, Monza
  - Piermarocchi Stefano, Padua
  - Neonatal Intensive Care Unit, Azienda Ospedaliera Universitaria Senese, Siena
  - Neonatal Intensive Care Unit, Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi, Varese

REFERENCES:
- [Background] Padrini L, Isacchi B, Bilia AR, Pini A, Lanzi C, Masini E, Della Bona ML, Calvani AM, Ceccantini R, la Marca G, Filippi L. Pharmacokinetics and local safety profile of propranolol eye drops in rabbits. Pediatr Res. 2014 Oct;76(4):378-85. doi: 10.1038/pr.2014.108. Epub 2014 Jul 16. PMID 25029260
- [Background] Filippi L, Cavallaro G, Bagnoli P, Dal Monte M, Fiorini P, Donzelli G, Tinelli F, Araimo G, Cristofori G, la Marca G, Della Bona ML, La Torre A, Fortunato P, Furlanetto S, Osnaghi S, Mosca F. Oral propranolol for retinopathy of prematurity: risks, safety concerns, and perspectives. J Pediatr. 2013 Dec;163(6):1570-1577.e6. doi: 10.1016/j.jpeds.2013.07.049. Epub 2013 Sep 18. PMID 24054431
- [Background] Dal Monte M, Casini G, la Marca G, Isacchi B, Filippi L, Bagnoli P. Eye drop propranolol administration promotes the recovery of oxygen-induced retinopathy in mice. Exp Eye Res. 2013 Jun;111:27-35. doi: 10.1016/j.exer.2013.03.013. Epub 2013 Mar 23. PMID 23528535
- [Background] Filippi L, Cavallaro G, Fiorini P, Malvagia S, Della Bona ML, Giocaliere E, Bagnoli P, Dal Monte M, Mosca F, Donzelli G, la Marca G. Propranolol concentrations after oral administration in term and preterm neonates. J Matern Fetal Neonatal Med. 2013 May;26(8):833-40. doi: 10.3109/14767058.2012.755169. Epub 2013 Jan 31. PMID 23205867
- [Background] Della Bona ML, Malvagia S, Villanelli F, Giocaliere E, Ombrone D, Funghini S, Filippi L, Cavallaro G, Bagnoli P, Guerrini R, la Marca G. A rapid liquid chromatography tandem mass spectrometry-based method for measuring propranolol on dried blood spots. J Pharm Biomed Anal. 2013 May 5;78-79:34-8. doi: 10.1016/j.jpba.2013.01.034. Epub 2013 Feb 4. PMID 23434527
- [Derived] Filippi L, Cavallaro G, Berti E, Padrini L, Araimo G, Regiroli G, Raffaeli G, Bozzetti V, Tagliabue P, Tomasini B, Mori A, Buonocore G, Agosti M, Bossi A, Chirico G, Aversa S, Fortunato P, Osnaghi S, Cavallotti B, Suzani M, Vanni M, Borsari G, Donati S, Nascimbeni G, Nardo D, Piermarocchi S, la Marca G, Forni G, Milani S, Cortinovis I, Calvani M, Bagnoli P, Dal Monte M, Calvani AM, Pugi A, Villamor E, Donzelli G, Mosca F. Propranolol 0.2% Eye Micro-Drops for Retinopathy of Prematurity: A Prospective Phase IIB Study. Front Pediatr. 2019 May 7;7:180. doi: 10.3389/fped.2019.00180. eCollection 2019. PMID 31134171
- [Derived] Filippi L, Cavallaro G, Berti E, Padrini L, Araimo G, Regiroli G, Bozzetti V, De Angelis C, Tagliabue P, Tomasini B, Buonocore G, Agosti M, Bossi A, Chirico G, Aversa S, Pasqualetti R, Fortunato P, Osnaghi S, Cavallotti B, Vanni M, Borsari G, Donati S, Nascimbeni G, la Marca G, Forni G, Milani S, Cortinovis I, Bagnoli P, Dal Monte M, Calvani AM, Pugi A, Villamor E, Donzelli G, Mosca F. Study protocol: safety and efficacy of propranolol 0.2% eye drops in newborns with a precocious stage of retinopathy of prematurity (DROP-ROP-0.2%): a multicenter, open-label, single arm, phase II trial. BMC Pediatr. 2017 Jul 14;17(1):165. doi: 10.1186/s12887-017-0923-8. PMID 28709412